CLINICAL TRIAL: NCT01671787
Title: A Phase 1b Randomized, Open Label, Active-Controlled Study to Assess the Safety, Viral Kinetics, and Anti-HBV Activity of GS-7340 in Treatment-Naive Adults With Chronic Hepatitis B (CHB) Infection
Brief Title: A Phase 1b Study Assessing GS-7340 in Treatment-Naive Adults With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-320-0101
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2014-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; HBV; GS-7340; TDF; Tenofovir disoproxil fumarate; Gilead; Viread
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- GS-7340 8mg (Experimental): After Screening procedures, eligible subjects will be randomized 1:1:1:1:1 to receive either open-label GS-7340 8, 25, 40, or 120 mg (3 x 40 mg), or open-label TDF 300 mg for 28 days.
  Interventions: Drug: GS-7340
- GS-7340 25mg (Experimental): After Screening procedures, eligible subjects will be randomized 1:1:1:1:1 to receive either open-label GS-7340 8, 25, 40, or 120 mg (3 x 40 mg), or open-label TDF 300 mg for 28 days.
  Interventions: Drug: GS-7340
- GS-7340 40mg (Experimental): After Screening procedures, eligible subjects will be randomized 1:1:1:1:1 to receive either open-label GS-7340 8, 25, 40, or 120 mg (3 x 40 mg), or open-label TDF 300 mg for 28 days.
  Interventions: Drug: GS-7340
- GS-7340 120mg (Experimental): After Screening procedures, eligible subjects will be randomized 1:1:1:1:1 to receive either open-label GS-7340 8, 25, 40, or 120 mg (3 x 40 mg), or open-label TDF 300 mg for 28 days.
  Interventions: Drug: GS-7340
- Tenofovir disoproxil fumarate 300mg (Experimental): After Screening procedures, eligible subjects will be randomized 1:1:1:1:1 to receive either open-label GS-7340 8, 25, 40, or 120 mg (3 x 40 mg), or open-label TDF 300 mg for 28 days.
  Interventions: Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: GS-7340 — Subjects are randomized to receive one of four different doses of GS-7340 over 28 days of therapy.
  Arms: GS-7340 120mg; GS-7340 25mg; GS-7340 40mg; GS-7340 8mg
Drug: Tenofovir disoproxil fumarate — Subjects will receive 300mg of Tenofovir disoproxil fumarate (TDF) over 28 days of therapy
  Other Names: Viread
  Arms: Tenofovir disoproxil fumarate 300mg

SUMMARY:
This is an open-label study evaluating multiple doses of GS-7340 versus Tenofovir disoproxil fumarate (TDF).

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled study whose primary objective is to evaluate the safety and efficacy of several doses of GS-7340. This study will evaluate the safety, viral kinetics, and antiviral activity of 4 different doses of GS-7340 over 28 days of therapy. In addition, the study will evaluate the antiviral activity of an optimal dose of GS-7340 versus 300mg Tenofovir disoproxil fumarate (TDF) over 28 days of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 65 years of age
* Must have Screening plasma HBV DNA ≥ 2x10^3 IU/mL
* Must have chronic HBV infection for at least 6 months
* Must have estimated creatinine clearance (CLCr) ≥ 70 mL/min
* Not pregnant or nursing
* Women must be of non-childbearing potential OR of childbearing potential with confirmed negative pregnancy tests
* Consistent and correct use of recommended methods of birth control for men and women

Exclusion Criteria:

* Pregnant or lactating subjects
* Receipt of anti-HBV nucleoside/nucleotide therapy. Subjects who have failed prior Interferon treatment, greater than 6 months prior to screening, are permitted to participate in the study screening
* Known co-infection with HIV, hepatitis C virus (HCV) or hepatitis D virus (HDV)
* Presence of autoimmune disorders
* History of liver disease other than Hepatitis B
* History of Gilbert's Disease
* Any sign of decompensated liver disease
* Known or suspected cirrhosis
* Evidence of hepatocellular carcinoma
* Presence or history of cardiovascular disease, cardiomyopathy, and/or cardiac conduction abnormalities
* Electrolyte abnormalities
* History of treatment that permanently alters the gastric condition
* Alcohol or substance abuse
* History of bleeding diathesis
* Significant bone disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in serum hepatitis B virus (HBV) DNA | Up to Week 4
  Time-weighted average change from baseline through Week 4 (DAVG4) in serum HBV DNA (log10 IU/mL) for GS-7340 8-, 25-, 40 and 120-mg.

SECONDARY OUTCOMES:
Change in HBV DNA for tenofovir disoproxil fumarate (TDF) | Up to Week 4
  Comparing the short-term antiviral activity of GS-7340 with TDF 300mg. This is measured by time-weighted average change from baseline through Week 4 (DAVG4) in serum HBV DNA (log10 IU/mL) for TDF.
Change in HBV DNA of GS-7340 through 28 days of therapy | Up to week 4
  Time weighted change from baseline to day 29 (DAVG4) in serum HBV DNA (log10 IU/mL)
Pharmacokinetics (PK) of GS-7340 and/or tenofovir (TVF) following single and multiple doses of GS-7340 and TDF | Up to week 4
  GS-7340 and tenofovir (TFV) PK parameters in plasma will be calculated as applicable: Cmax, Tmax, Clast, Tlast, T1/2, λz, AUC0-t, AUC0-last, AUC0-∞, %AUCexp.
  PK samples are collected on:
  * Baseline/Day 1: 0 (predose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post dose
  * Additional predose plasma samples will be collected on Days 2, 5, 8, 10, 15, 19, 22, and 29/End of Treatment.
Safety and Tolerability of Therapy | Up to week 4
  Safety and tolerability is measured by the incidence of adverse events and graded laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, MD, Study Director — Gilead Sciences
Locations (19):
- United States (4):
  - Research and Education Inc., San Diego, California
  - University of Maryland Institute of Human Virology, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Baylor College of Medicine - St. Luke's Episcopal Hospital, Houston, Texas
- Australia (4):
  - Monash Medical Centre, Melborne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Canada (5):
  - Downtown Infectious Diseases Clinic (University of British Columbia), Vancouver, British Columbia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Algorithme Pharma, Montreal, Quebec
  - Pro-recherche, Saint Romuald, Quebec
- Auckland Clinical Studies, Auckland, New Zealand
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Grahame Hayton Unit, London
  - University College London Hospital, London
  - Institute of Liver Studies, King's College Hospital, London
  - Nottingham University Hospitals NHS Trust - Queens Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency